CLINICAL TRIAL: NCT02832856
Title: Testing the Effectiveness of the Full and Abridged Versions of the Relationship Smarts Curriculum for 9th Grade Students
Brief Title: Testing the Effectiveness of the Full and Abridged Relationship Smarts Curriculum for 9th Grade Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MPR-500098-MTC
Record Dates: First submitted 2016-07-08; First posted 2016-07-14 (Estimated); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Attitudes; Knowledge
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Placebo Comparator): Control group members will receive a job readiness curriculum entitled Beginning to Work it Out (BWIO) that assists at-risk youth who are preparing for first-time employment. Topics include recognizing how personal beliefs and behaviors may be perceived in the workplace, as well as "soft skills" such as emotional self-management and problem-solving skills.
  Interventions: Behavioral: Job Readiness Curriculum
- Full Relationship Smarts Curriculum (Experimental): This group receives the behavioral intervention of the healthy relationship education in the form of the full, 12-lesson RS+ curriculum over approximately 12 weeks.
  Interventions: Behavioral: Healthy Relationship Education
- Abridged Relationship Smarts Curriculum (Experimental): This group receives the behavioral intervention of the healthy relationship education in the form of the "summary" 8-lesson version of the RS+ curriculum - as well as four lessons on career planning and job readiness over approximately 12 weeks.
  Interventions: Behavioral: Healthy Relationship Education; Behavioral: Job Readiness Curriculum

INTERVENTIONS:
Behavioral: Healthy Relationship Education — RS+ is a widely-implemented healthy relationship education curriculum that aligns with the Georgia Department of Education performance standards in health education. The full curriculum features 12 lessons covering such topics as healthy relationships, dating violence prevention, communication skills, conflict management, and decision making.
  Arms: Abridged Relationship Smarts Curriculum; Full Relationship Smarts Curriculum
Behavioral: Job Readiness Curriculum — Beginning to Work it Out (BWIO) assists youth who are preparing for first-time employment. Topics include recognizing how personal beliefs and behaviors may be perceived in the workplace, as well as "soft skills" such as emotional self-management and problem-solving skills.
  Arms: Abridged Relationship Smarts Curriculum; Control

SUMMARY:
This evaluation will test the program effectiveness of a relationship education program (Relationship Smarts PLUS)and an abridged version of the program to 9th Grade Students on outcomes of knowledge. It will test 1) whether the Relationship Smarts (RS) Curriculum is more effective than a control curriculum of job-readiness programming, and 2) whether an abridged 8-lesson version of the RS Curriculum can be as effective as the full 12-lesson version.

DETAILED DESCRIPTION:
MTCI plans to deliver the Relationship Smarts PLUS (RS+) education curriculum to youth in high schools during the regular school day. RS+ is a widely-implemented healthy relationship education curriculum that aligns with the Georgia Department of Education performance standards in health education. The curriculum features 12 lessons covering such topics as healthy relationships, dating violence prevention, communication skills, conflict management, and decision making. MORE THAN CONQUERORS, INC. (MTCI) plans to deliver the curriculum to 9th grade students as part of a required, semester-long health class. The program will be delivered by trained facilitators from MTCI in coordination with each participating school.

To be eligible to participate, students must be enrolled in one of the targeted health classes and have permission from a parent or guardian to participate in both the MATURE Plus II program and the STREAMS evaluation.The study plans to enroll 1,840 students over the entire two-year evaluation period.

At the start of each semester, the targeted sections of 9th grade health class will be randomly assigned into one of three research groups: (1) a group that receives the full, 12-lesson RS+ curriculum, (2) a group that receives a "summary" 8-lesson version of the RS+ curriculum and four lessons on career planning and job readiness, or (3) a control group that receives lessons on career planning and job readiness without any lessons from the RS+ curriculum.

All students for whom consent and assent have been obtained will be asked to complete three surveys: (1) a baseline survey administered in health class near the start of the semester, (2) a post-program survey administered in health class near the end of the semester, and (3) a one-year follow-up survey administered about 12 months after the baseline survey, during 10th grade

ELIGIBILITY:
Inclusion Criteria:

* high school students in 9th grade health classes
* must be enrolled in one of the targeted health classes
* permission from a parent or guardian to participate in both the program and the evaluation

Exclusion Criteria:

* non-students
* students in other grades of high school
* students not enrolled in health class
* students without parental permission to participate

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1180 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Perceived general relationship skills | one year after random assignment
  Six-item scale (range: 1 to 4)
Perceived conflict management skills | one year after random assignment
  Five-item scale (range: 1 to 4)
Disapproval of teen dating violence | one year after random assignment
  Twelve-item scale (range: 1 to 4)
Constraining beliefs about marriage | one year after random assignment
  Series of three separate continuous variables (range: 1 to 4)
Knowledge of pregnancy and STIs | one year after random assignment
  Continuous index variable: sum of correct responses to five true/false statements
Desire to avoid teen pregnancy | one year after random assignment
  series of three separate continuous variables (range: 1 to 4)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Goesling, PhD, Principal Investigator — Mathematica Policy Research
Locations (1):
- More Than Conquerors, Inc., Conyers, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Restricted use files will be made available to researchers through the Inter-University Consortium for Political and Social Research (ICPSR) at the University of Michigan
Time Frame: Mid-2022
Access Criteria: Yet to be determined.